CLINICAL TRIAL: NCT07027891
Title: ROMIAE 2 Trial: Randomized Controlled Trial for Managing Suspicious Acute Myocardial Infarction in ED Using AI-ECG
Brief Title: The Rule-Out Acute Myocardial Infarction Using Aritifical Intelligence Electrocardiogram (ROMIAE) 2 Trial
Acronym: ROMIAE 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Kyuseok Kim, Professor, MD, PhD, CHA University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ROMIAE II trial; RS-2025-02213791 (Other Grant/Funding Number: Korea Health Technology R&D Project)
Record Dates: First submitted 2025-05-27; First posted 2025-06-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction (MI); Chest Pain Rule Out Myocardial Infarction
Keywords: chest pain, suspicious myocardial infarction; artificial intelligence; electrocardiogram; emergency department; acute coronary syndrome; AI/ML-enabled SaMd
MeSH Terms: conditions — Myocardial Infarction; Chest Pain; Emergencies; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The patients in control group would be managed with usual care using HEART score in addition to recent acute coronary syndrome guideline.
- AI-ECG group (Experimental): The patients in AI-ECG group would be managed with the information of the myocardial infarction risk score in AI-ECG in addition to the usual care.
  Interventions: Device: AI-ECG

INTERVENTIONS:
Device: AI-ECG — The patients in AI-ECG group would be managed with the information of the myocardial infarction risk score in AI-ECG in addition to the usual care.
  Arms: AI-ECG group

SUMMARY:
This study is to see whether the AI ECG assisted protocol is as safe and efficacious as conventional protocol in early triage of suspected myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* chest pain
* suspicious of acute myocardial infarction

Exclusion Criteria:

* STEMI
* Revisit of same symptoms within 1 week
* traumatic chest pain
* Pneumothorax
* Transferred from other hospital diagnosed of AMI
* Cardiac arrest
* Chest pain of clearly non-cardiac etiology
* declined to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4670 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
30 Days MACE(Major adverse cardiac events) | 30 days
  Death, acute myocardial infarction, stroke, target vessel revascularization, stent thrombosis within 30 days from index visit

SECONDARY OUTCOMES:
Missed acute myocardial infarction at index visit | 30 days
  Missed acute myocardial infarction at index ED visit, but is detected later in anyplace (Outpatient clinic, revisit to ED, or other hospital, etc)
AI-ECG 30 days MACE prediction performance | 30 days
  AUROC and AUPRC by continuous AI-ECG score
AI-ECG 30 days MACE prediction performance | 30 Days
  Sensitivity and specificity by pre-specified cutoff thresholds for Low to intermediate risk or intermediate to high risk
AI-ECG 30 days MACE prediction performance | 30 Days
  Positive predictive value and Negative predictive value by pre-specified cutoff thresholds for Low to intermediate risk or intermediate to high risk
AI-ECG acute myocardial infarction (index visit) discrimination performance | 30 days
  AUROC and AUPRC by continuous AI-ECG score
AI-ECG acute myocardial infarction (index visit) discrimination performance | 30 Days
  Sensitivity and Specificity by pre-specified cutoff thresholds for Low to intermediate risk or intermediate to high risk
AI-ECG acute myocardial infarction (index visit) discrimination performance | 30 Days
  Positive predictive value and Negative predictive value by pre-specified cutoff thresholds for Low to intermediate risk or intermediate to high risk
Medical resources utilization | 30 days
  Length of stay in ED
Medical resources utilization | 24 hours
  early discharge from ED(within 4 hours)
Medical resources utilization | 7 Days
  Revisit to ED with same symptoms within 1 week
Medical resources utilization | 30 days
  Admission rate
Medical resources utilization | 30 days
  length of stay in hospital
Medical resources utilization | 30 days
  It would be evaluated by the rate of all additional tests including cardiac CT, coronary angiography, echocardiography, and stress test.
Medical resources utilization | 30 days
  Direct medical cost

OTHER OUTCOMES:
Compliance of medical doctor in AI-ECG low risk group | 7 days
  Compliance of medical doctors to AI-ECG results in AI-ECG low risk group according to the study period(Q1 to Q4), which would be evaluated by discharge rate from ED.
Compliance of medical doctor in AI-ECG low risk group | 7 days
  Compliance of medical doctors to AI-ECG results in AI-ECG low risk group according to the study period(Q1 to Q4), which would be evaluated by the rate of no follow-up troponin check.
Compliance of medical doctor in AI-ECG low risk group | 7 days
  Compliance of medical doctors to AI-ECG results in AI-ECG low risk group according to the study period(Q1 to Q4), which would be evaluated by the rate of only baseline and 1 h follow-up troponin check
Compliance of medical doctor in AI-ECG high risk group | 7 Days
  Compliance of medical doctors to AI-ECG results in AI-ECG high risk group according to the study period(Q1 to Q4), which would be evaluated by admission rate.
Compliance of medical doctor in AI-ECG high risk group | 7 Days
  Compliance of medical doctors to AI-ECG results in AI-ECG high risk group according to the study period(Q1 to Q4), which would be evaluated by the sum rate of additional tests such as coronary artery CT, CAG, stress test.
Compliance of medical doctor in AI-ECG high risk group | 7 Days
  Compliance of medical doctors to AI-ECG results in AI-ECG high risk group according to the study period(Q1 to Q4), which would be evaluated by the rate of full check up of troponin(0, 1h, 2h).
Compliance of medical doctor in AI-ECG high risk group | 7 Days
  Compliance of medical doctors to AI-ECG results in AI-ECG high risk group according to the study period(Q1 to Q4), which would be evaluated by time from ED to admission.
Compliance of medical doctor in AI-ECG high risk group | 7 Days
  Compliance of medical doctors to AI-ECG results in AI-ECG high risk group according to the study period(Q1 to Q4), which would be evaluated by time to CAG.
Compliance of medical doctor in AI-ECG high risk group | 7 Days
  Compliance of medical doctors to AI-ECG results in AI-ECG high risk group according to the study period(Q1 to Q4), which would be evaluated by cardiology contact rate.
Satisfaction score of patients | 7 Days
  Satisfaction score using AI-ECG from 1-10 (1 is lowest, 10 is highest)
Satisfaction score of medical personnel | 7 Days
  Satisfaction score using AI-ECG from 1-10 (1 is lowest, 10 is highest)
AI-ECG occlusive myocardial infarction detection performance | 30 days
  AUROC and AUPRC by continuous AI-ECG score
AI-ECG occlusive myocardial infarction detection performance | 30 days
  Sensitivity and Specificity by pre-specified cutoff thresholds for Low to intermediate risk or intermediate to high risk
AI-ECG occlusive myocardial infarction detection performance | 30 days
  Positive predictive value and Negative predictive value by pre-specified cutoff thresholds for Low to intermediate risk or intermediate to high risk

CONTACTS AND LOCATIONS:
Overall Officials: KYUSEOK Kim, MD, PhD, Principal Investigator — CHA University
Locations (12):
- South Korea (12):
  - Asan Medical Center, Seoul
  - CHA Bundang Medical Center, Seoul
  - Ewha Womans University, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hanyang University, Seoul
  - Jeonbuk National University Hospital, Seoul
  - Korea University Ansan Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Soonchunhyang University Bucheon Hospital, Seoul
  - Yonsei University Wonju College of Medicine, Seoul

IPD SHARING:
Plan to Share IPD: Yes
The data would be shared with other researchers when they contact to the principal investigator with reasonable context.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code